CLINICAL TRIAL: NCT06141473
Title: Master Protocol of Two Independent, Randomized, Double-blind, Phase 3 Studies Comparing Efficacy and Safety of Frexalimab (SAR441344) to Teriflunomide in Adult Participants With Relapsing Forms of Multiple Sclerosis
Brief Title: Efficacy and Safety Studies of Frexalimab (SAR441344) in Adults With Relapsing Forms of Multiple Sclerosis
Acronym: FREXALT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17919; 2023-504358-36 (Registry Identifier: CTIS); U1111-1290-9326 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide; Cholestyramine Resin; Charcoal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Frexalimab (Experimental): Participants will receive Frexalimab infusion and placebo tablet.
  Interventions: Drug: Frexalimab; Drug: Placebo tablet; Drug: MRI contrast-enhancing agents; Drug: Cholestyramine; Drug: Activated charcoal
- Teriflunomide (Active Comparator): Participants will receive teriflunomide tablet and placebo infusion.
  Interventions: Drug: Teriflunomide; Drug: Placebo infusion; Drug: MRI contrast-enhancing agents; Drug: Cholestyramine; Drug: Activated charcoal

INTERVENTIONS:
Drug: Frexalimab — SAR441344 Solution for IV infusion
  Arms: Frexalimab
Drug: Teriflunomide — Aubagio oral tablet
  Arms: Teriflunomide
Drug: Placebo infusion — Solution for IV infusion
  Arms: Teriflunomide
Drug: Placebo tablet — Oral tablet
  Arms: Frexalimab
Drug: MRI contrast-enhancing agents — IV, as per respective label
Drug: Cholestyramine — oral, 8 g 3 times daily for 11 days for accelerated elimination procedure (4 g 3 times daily for 11 days in case of intolerance). The teriflunomide local label should be followed.
Drug: Activated charcoal — oral, 50 g every 12 hours for 11 days for accelerated elimination procedure. The teriflunomide local label should be followed.

SUMMARY:
The purpose of each study is to independently measure the annualized relapse rate (ARR) with administration of frexalimab compared to a daily oral dose of teriflunomide in male and female participants with relapsing forms of multiple sclerosis (aged 18 to 55 years at the time of enrollment). People diagnosed with relapsing forms of multiple sclerosis are eligible for enrollment as long as they meet all the inclusion criteria and none of the exclusion criteria.

Study details include:

* This event-driven study will have variable duration depending on the recruitment rate, the event rate, the study discontinuation rate and the 12-month minimum treatment duration. Different participants will have different study durations. The last participant randomized will have at least 12 months of study duration, and assuming a 28-month recruitment period, the first participant randomized will have 40 months or longer of study duration.
* The study intervention duration will vary similarly as the study duration.
* The assessment of scheduled visits will include 1 common end of study [EOS] visit and 3 follow-up visits) with a visit frequency of every 4 weeks for the first 6 months and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have been diagnosed with RMS according to the 2017 revision of the McDonald diagnostic criteria.
* The participant has an EDSS score ≤5.5 at the first visit (Screening Visit)
* The participant must have at least 1 of the following prior to screening:

  * ≥1 documented relapse within the previous year OR
  * ≥2 documented relapses within the previous 2 years, OR
  * ≥1 documented Gd enhancing lesion on an MRI scan within the previous year.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* The participant has been diagnosed with PPMS according to the 2017 revision of the McDonald diagnostic criteria
* The participant has a history of infection or may be at risk for infection:
* The presence of psychiatric disturbance or substance abuse.
* History, clinical evidence, suspicion or significant risk for thromboembolic events, as well as myocardial infarction, stroke, and/or antiphosholipid syndrome and any participants requiring antithrombotic treatment.
* Current hypogammaglobulinemia defined by Ig levels below the LLN at Screening or a history of primary hypogammaglobulinemia.
* A history or presence of disease that can mimic MS symptoms, such as, but not limited to neuromyelitis optica spectrum disorder, systemic lupus erythematosus, Sjogren's syndrome, acute disseminated encephalomyelitis, and myasthenia gravis.
* The participant has had a relapse in the 30 days prior to randomization.
* The participant has contraindication for MRI, ie, presence of pacemaker, metallic implants in high risk areas (ie, artificial heart valves, aneurysm/vessel clips), presence of metallic material (eg, shrapnel) in high risk areas, known history of allergy to any contrast medium, or history of claustrophobia that would prevent completion of all protocol scheduled MRI scans.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-05-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate (ARR) during the study period assessed by protocol defined adjudicated relapses | Until Week 156
  ARR during the study period assessed by protocol-defined adjudicated relapses. This endpoint will be analyzed in the ITT population of each study using a negative binomial model with the total number of adjudicated relapses per participant occurring during the observation period as the response variable and with terms for treatment group, Gd-enhancing T1 lesions at baseline (presence, absence), EDSS strata (<4, ≥4), and geographical region (US, non-US).

SECONDARY OUTCOMES:
Time to onset of composite confirmed disability worsening (cCDW) | Until Week 156
  confirmed over 6 months as assessed by the composite of:
  * increase from the baseline expanded disability status scale (EDSS) score of ≥1.5 points when the baseline is 0, or ≥1.0 point when the baseline is 0.5 to 5.0, or ≥0.5 point when the baseline is ≥5.5, OR
  * increase of ≥20% from the baseline time in the 9-hole peg test (9HPT), OR
  * increase of ≥20% from the baseline time in the Timed 25-foot walk (T25FW) test
Time to onset of cCDW, confirmed over 3 months | Until Week 156
Time to onset of individual components of the composite, confirmed over 3-months or 6-months | Until Week 156
Time to onset of confirmed disability improvement (CDI) | Until Week 156
  defined as decrease from baseline EDSS score of ≥1.0 or ≥ 0.5 points when the baseline is ≥2 to ≤5.5 or >5.5 points, respectively, confirmed over 6 months. No improvement possible for 0 to 1.5 points
Progression independent of relapse activity defined as the time to onset of 6-month cCDW | Until Week 156
  defined by either no prior relapse or an onset more than 90 days after the start date of the last investigatorreported relapse
Total number of new and/or enlarging T2 hyperintense lesions as detected by MRI | Until Week 156
  defined as the sum of the individual number of new and/or enlarging T2 lesions at all scheduled visits starting after baseline up to and including the EOS visit
Total number of new Gd-enhancing T1hyperintense lesions per scan as detected by MRI | Until Week 156
  defined as the sum of the individual number of new Gd enhancing T1-hyperintense lesions at all scheduled visits starting after baseline up to and including the EOS visit divided by the number of scans
Percent change in brain volume loss as detected by brain MRI scans at the EOS compared to Month 6 | From Week 24 to Week 156
Change in cognitive function at the EOS compared to baseline as assessed by the symbol digit modalities test (SDMT) | From baseline to Week 156
Change from baseline in multiple sclerosis impact scale 29 version 2 (MSIS-29v2) questionnaire scores over time | From baseline to Week 156
Change from baseline in patient reported outcome measurement information system (PROMIS) Fatigue MS-8 over time | Until Week 156
Number of participants with adverse events, SAEs, AEs leading to permanent study intervention discontinuation, AESIs and safety scales during the study period | Until Week 168
Number of participants with potentially clinically significant abnormality (PCSAs) in laboratory tests, ECG and vital signs during the study period | Until Week 168
  12-lead ECG (electrocardiogram) will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Number of participants with antidrug (ADAs) over time | Until Week 156
Change from baseline in plasma neurofilament light chain (NfL) levels over time | Until Week 144
Frexalimab plasma concentration over time | Until Week 144

CONTACTS AND LOCATIONS:
Locations (385):
- United States (100):
  - Alabama Neurology Associates- Site Number : 8400115, Birmingham, Alabama
  - The University of Alabama at Birmingham- Site Number : 8401135, Birmingham, Alabama
  - ~North Central Neurology Associates, PC- Site Number : 8401100, Cullman, Alabama
  - Dignity Health St. Joseph's Hospital and Medical Center- Site Number : 8401139, Phoenix, Arizona
  - Perseverance Research Center, LLC- Site Number : 8401138, Scottsdale, Arizona
  - Clinical Endpoints- Site Number : 8400050, Scottsdale, Arizona
  - The Research Center of Southern California, LLC- Site Number : 8400023, Carlsbad, California
  - University of California, Irvine- Site Number : 8401143, Irvine, California
  - Multiple Sclerosis Center of California- Site Number : 8401122, Laguna Hills, California
  - Chemidox Clinical Trials Inc.- Site Number : 8401157, Lancaster, California
  - Hoag Memorial Hospital- Site Number : 8401031, Newport Beach, California
  - Regina Berkovich, MD, PhD- Site Number : 8400005, West Hollywood, California
  - University of Colorado Health Science Center- Site Number : 8401001, Aurora, Colorado
  - Advanced Neurosciences Research- Site Number : 8401148, Fort Collins, Colorado
  - Hartford Healthcare Medical Group- Site Number : 8401069, Norwich, Connecticut
  - New England Institute for Clinical Research- Site Number : 8400114, Stamford, Connecticut
  - Georgetown University Hospital- Site Number : 8400044, Washington D.C., District of Columbia
  - Neurology of Central Florida Research Center, LLC- Site Number : 8401147, Altamonte Springs, Florida
  - Neurology Offices of South Florida- Site Number : 8401169, Boca Raton, Florida
  - First Choice Neurology - Espinosa Neurosciences- Site Number : 8401071, Boca Raton, Florida
  - Nova Clinical Research, LLC- Site Number : 8400189, Bradenton, Florida
  - Mayo Clinic- Site Number : 8401093, Jacksonville, Florida
  - Neurology Associates, PA- Site Number : 8400010, Maitland, Florida
  - University of Miami- Site Number : 8401177, Miami, Florida
  - Research by Design, LLC- Site Number : 8401191, Miami Lakes, Florida
  - Orlando Health Neuroscience Institute- Site Number : 8400060, Orlando, Florida
  - Axiom Clinical Research of Florida- Site Number : 8400049, Tampa, Florida
  - University of South Florida- Site Number : 8400013, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology- Site Number : 8401105, West Palm Beach, Florida
  - Savannah Neurology Specialists- Site Number : 8400061, Savannah, Georgia
  - Joi Life Wellness Group LLC- Site Number : 8401192, Smyrna, Georgia
  - NorthShore University Healthsystem- Site Number : 8401111, Evanston, Illinois
  - Consultants In Neurology- Site Number : 8401020, Northbrook, Illinois
  - Springfield Clinic, LLP- Site Number : 8400043, Springfield, Illinois
  - Indiana University Health, Inc- Site Number : 8400058, Fort Wayne, Indiana
  - Neuroscience Institute Center- Site Number : 8400053, Merrillville, Indiana
  - University Of Iowa Hospitals And Clinics- Site Number : 8400029, Iowa City, Iowa
  - University of Kansas Medical Center- Site Number : 8400084, Kansas City, Kansas
  - KC Research Center- Site Number : 8400032, Roeland Park, Kansas
  - Baptist Health Lexington- Site Number : 8401149, Lexington, Kentucky
  - Norton Neurology MS Services- Site Number : 8401103, Louisville, Kentucky
  - Neuromedical Clinic of CENLA, LLC- Site Number : 8401159, Alexandria, Louisiana
  - DelRicht Research- Site Number : 8401182, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation- Site Number : 8400027, New Orleans, Louisiana
  - International Neurorehabilitation Institute- Site Number : 8400089, Lutherville, Maryland
  - Boston Clinical Trials- Site Number : 8401178, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center- Site Number : 8401041, Boston, Massachusetts
  - Neurology Center of New England PC- Site Number : 8401164, Foxborough, Massachusetts
  - ~Henry Ford Hospital- Site Number : 8401091, Detroit, Michigan
  - Michigan Institute For Neurological Disorders- Site Number : 8400004, Farmington Hills, Michigan
  - Trinity Health Grand Rapids- Site Number : 8400150, Grand Rapids, Michigan
  - Memorial Healthcare Institute for Neuroscience- Site Number : 8400123, Owosso, Michigan
  - Profound Research / Rochester Medical Group / Michigan Health Partners- Site Number : 8401172, Rochester Hills, Michigan
  - University of Minnesota- Site Number : 8400056, Minneapolis, Minnesota
  - Minnesota Center for Multiple Sclerosis- Site Number : 8400073, Plymouth, Minnesota
  - Sharlin Health & Neurology- Site Number : 8400016, Ozark, Missouri
  - Washington University School of Medicine- Site Number : 8400076, St Louis, Missouri
  - The MS Center for Innovations in Care- Site Number : 8401141, St Louis, Missouri
  - Lou Ruvo Center for Brain Health- Site Number : 8400045, Las Vegas, Nevada
  - Renown Institute for Neurosciences- Site Number : 8400066, Reno, Nevada
  - Rutgers University - Robert Wood Johnson Medical School- Site Number : 8401067, New Brunswick, New Jersey
  - University of New Mexico- Site Number : 8401090, Albuquerque, New Mexico
  - NYU Langone South Shore Neurologic Associates- Site Number : 8400063, Patchogue, New York
  - Montefiore Medical Center- Site Number : 8401145, The Bronx, New York
  - The Neurological Institute, PA- Site Number : 8401166, Charlotte, North Carolina
  - Piedmont Healthcare/Research- Site Number : 8400002, Charlotte, North Carolina
  - Velocity Clinical Research, Inc- Site Number : 8400014, Raleigh, North Carolina
  - Atrium Health Wake Forest Baptist- Site Number : 8400040, Winston-Salem, North Carolina
  - Sanford Brain and Spine Center- Site Number : 8401085, Fargo, North Dakota
  - Dayton Center for Neurological Disorders- Site Number : 8400079, Centerville, Ohio
  - University of Cincinnati Medical Center- Site Number : 8401117, Cincinnati, Ohio
  - Ohio State University- Site Number : 8401009, Columbus, Ohio
  - Ohio Health Research Institute- Site Number : 8401092, Columbus, Ohio
  - The Boster Center for Multiple Sclerosis- Site Number : 8400006, Columbus, Ohio
  - University of Cincinnati- Site Number : 8401008, Dayton, Ohio
  - Oklahoma Medical Research Foundation- Site Number : 8400039, Oklahoma City, Oklahoma
  - Providence Multiple Sclerosis Center- Site Number : 8400052, Portland, Oregon
  - Oregon Neurology- Site Number : 8400188, Springfield, Oregon
  - Abington Neurological Associates- Site Number : 8401065, Abington, Pennsylvania
  - Penn State University Milton S. Hershey Medical Center- Site Number : 8401176, Hershey, Pennsylvania
  - Comprehensive MS Center Thomas Jefferson University Hospital- Site Number : 8400035, Philadelphia, Pennsylvania
  - Allegheny Health Network- Site Number : 8401173, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital- Site Number : 8401133, Pittsburgh, Pennsylvania
  - Premier Neurology- Site Number : 8401047, Greenville, South Carolina
  - HOPE Neurology- Site Number : 8400019, Knoxville, Tennessee
  - Neurology Consultants of Dallas- Site Number : 8400152, Dallas, Texas
  - ANESC Research- Site Number : 8400187, El Paso, Texas
  - Baylor College of Medicine (BCM) Ad Board- Site Number : 8401170, Houston, Texas
  - North Texas Institute of Neurology - Plano- Site Number : 8401083, Plano, Texas
  - UTHSCSA- Site Number : 8401167, San Antonio, Texas
  - Lone Star Neurology of San Antonio- Site Number : 8400099, San Antonio, Texas
  - Texas Institute for Neurological Disorders-Sherman- Site Number : 8400018, Sherman, Texas
  - INOVA Neurology- Site Number : 8401109, Fairfax, Virginia
  - MS Center of Greater Washington- Site Number : 8401128, Vienna, Virginia
  - Sentara Neurological Associates- Site Number : 8401168, Virginia Beach, Virginia
  - Multiple Sclerosis Center, Swedish Neuroscience Institute- Site Number : 8400078, Seattle, Washington
  - University of Washington MS Center- Site Number : 8401146, Seattle, Washington
  - MultiCare Neuroscience Center of Washington- Site Number : 8401140, Tacoma, Washington
  - Wheaton Franciscan Healthcare- Site Number : 8400034, Milwaukee, Wisconsin
  - Medical College of Wisconsin- Site Number : 8400038, Milwaukee, Wisconsin
- Argentina (7):
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320008, CABA, Buenos Aires
  - Investigational Site Number : 0321010, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320009, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320001, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0321011, Córdoba, Córdoba Province
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
- Austria (3):
  - Investigational Site Number : 0400001, Innsbruck
  - Investigational Site Number : 0401002, Linz
  - Investigational Site Number : 0401003, Vienna
- Belgium (2):
  - Investigational Site Number : 0560006, Ghent
  - Investigational Site Number : 0560005, Overpelt
- Brazil (17):
  - CEDOES - Centro de Diagnostico e Pesquisa de Osteoporose do ES- Site Number : 0761029, Vitória, Espírito Santo
  - Instituto Bahiano de Imunoterapia - IBIS- Site Number : 0761030, Salvador, Estado de Bahia
  - Clinica AMO- Site Number : 0761017, Salvador, Estado de Bahia
  - L2IP Instituto de Pesquisas Clinicas- Site Number : 0760003, Brasília, Federal District
  - HC UFG - Hospital Das Clinicas de Goias- Site Number : 0761024, Goiânia, Goiás
  - Freire Pesquisa Clínica- Site Number : 0761025, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba- Site Number : 0761001, Curitiba, Paraná
  - Hospital Moinhos de Vento - HMV - Site Number : 0761005, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Neurológica- Site Number : 0761031, Porto Alegre, Rio Grande do Sul
  - Instituto Ceos- Site Number : 0761028, Porto Alegre, Rio Grande do Sul
  - Instituto do Cerebro - InsCer- Site Number : 0761009, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica e Neurocirurgica de Joinville - NEUROLOGICA- Site Number : 0761007, Joinville, Santa Catarina
  - Hospital Christovao Da Gama- Site Number : 0761022, Santo André, São Paulo
  - CPQuali Pesquisa Clinica- Site Number : 0761002, São Paulo, São Paulo
  - PSEG Centro de Pesquisa Clinica- Site Number : 0761021, São Paulo, São Paulo
  - Centro Medico Sinapse- Site Number : 0761004, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas- Site Number : 0761027, São Paulo
- Bulgaria (9):
  - Investigational Site Number : 1000009, Blagoevgrad
  - Investigational Site Number : 1001008, Panagyurishte
  - Investigational Site Number : 1000007, Pazardzhik
  - Investigational Site Number : 1001010, Pleven
  - Investigational Site Number : 1000002, Pleven
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1001001, Sofia
  - Investigational Site Number : 1001006, Sofia
  - Investigational Site Number : 1000005, Sofia
- Canada (9):
  - Investigational Site Number : 1240017, Edmonton, Alberta
  - Investigational Site Number : 1240010, Vancouver, British Columbia
  - Investigational Site Number : 1240007, St. John's, Newfoundland and Labrador
  - Investigational Site Number : 1240014, London, Ontario
  - Investigational Site Number : 1240002, Ottawa, Ontario
  - Investigational Site Number : 1240001, Gatineau, Quebec
  - Investigational Site Number : 1240004, Granby, Quebec
  - Investigational Site Number : 1240008, Lévis, Quebec
  - Investigational Site Number : 1240003, Québec
- Chile (5):
  - Investigational Site Number : 1521005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1521001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1521003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago
- China (29):
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560008, Beijing
  - Investigational Site Number : 1560007, Beijing
  - Investigational Site Number : 1560003, Changchun
  - Investigational Site Number : 1560011, Changsha
  - Investigational Site Number : 1560004, Chengdu
  - Investigational Site Number : 1561029, Chengdu
  - Investigational Site Number : 1560015, Chongqing
  - Investigational Site Number : 1560020, Dongguan
  - Investigational Site Number : 1561028, Fuzhou
  - Investigational Site Number : 1561026, Guangzhou
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1561023, Hangzhou
  - Investigational Site Number : 1561027, Harbin
  - Investigational Site Number : 1560040, Hohhot
  - Investigational Site Number : 1560019, Hohhot
  - Investigational Site Number : 1561025, Jinan
  - Investigational Site Number : 1560018, Nanjing
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560043, Shanghai
  - Investigational Site Number : 1560014, Shenyang
  - Investigational Site Number : 1560010, Shijiazhuang
  - Investigational Site Number : 1560030, Suzhou
  - Investigational Site Number : 1560006, Taiyuan
  - Investigational Site Number : 1560012, Tianjin
  - Investigational Site Number : 1560016, Wenzhou
  - Investigational Site Number : 1560009, Wuhan
  - Investigational Site Number : 1560013, Xi'an
  - Investigational Site Number : 1560021, Yinchuan
- Investigational Site Number : 1911001, Zagreb, Croatia
- Czechia (11):
  - Investigational Site Number : 2031011, Brno
  - Investigational Site Number : 2030005, Brno
  - Investigational Site Number : 2030002, Hradec Králové
  - Investigational Site Number : 2030006, Jihlava
  - Investigational Site Number : 2031007, Ostrava - Poruba
  - Investigational Site Number : 2030010, Pardubice
  - Investigational Site Number : 2031003, Prague
  - Investigational Site Number : 2031004, Prague
  - Investigational Site Number : 2031008, Praha 5 - Motol
  - Investigational Site Number : 2031009, Teplice
  - Investigational Site Number : 2030001, Zlín
- Denmark (2):
  - Investigational Site Number : 2081002, Esbjerg
  - Investigational Site Number : 2081001, Glostrup Municipality
- France (6):
  - Investigational Site Number : 2501017, Calais
  - Investigational Site Number : 2501018, Colmar
  - Investigational Site Number : 2501006, Grenoble
  - Investigational Site Number : 2501009, Lille
  - Investigational Site Number : 2501002, Nice
  - Investigational Site Number : 2501010, Saint-Herblain
- Germany (13):
  - Investigational Site Number : 2761014, Berlin
  - Investigational Site Number : 2761009, Bielefeld
  - Investigational Site Number : 2760010, Bochum
  - Investigational Site Number : 2761016, Böblingen
  - Investigational Site Number : 2760012, Dresden
  - Investigational Site Number : 2760002, Düsseldorf
  - Investigational Site Number : 2761013, Erbach im Odenwald
  - Investigational Site Number : 2761011, Essen
  - Investigational Site Number : 2761007, Jena
  - Investigational Site Number : 2760003, Leipzig
  - Investigational Site Number : 2761008, Marburg
  - Investigational Site Number : 2761006, Münster
  - Investigational Site Number : 2760001, Ulm
- Greece (5):
  - Investigational Site Number : 3001005, Athens
  - Investigational Site Number : 3000004, Ioannina
  - Investigational Site Number : 3001001, Larissa
  - Investigational Site Number : 3000002, Thessaloniki
  - Investigational Site Number : 3001006, Thessaloniki
- Investigational Site Number : 3441001, Shatin, Hong Kong
- Hungary (5):
  - Investigational Site Number : 3481003, Budapest
  - Investigational Site Number : 3481004, Budapest
  - Investigational Site Number : 3480002, Győr
  - Investigational Site Number : 3480001, Kaposvár
  - Investigational Site Number : 3481005, Pécs
- India (10):
  - Investigational Site Number : 3561024, Bengaluru
  - Investigational Site Number : 3560002, Chandigarh
  - Investigational Site Number : 3560017, Delhi
  - Investigational Site Number : 3560020, Kochi
  - Investigational Site Number : 3560010, Nagpur
  - Investigational Site Number : 3561005, Nashik
  - Investigational Site Number : 3561023, New Delhi
  - Investigational Site Number : 3561008, Punjagutta
  - Investigational Site Number : 3561006, Shimla
  - Investigational Site Number : 3561004, Thiruvananthapuram
- Israel (3):
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760002, Safed
  - Investigational Site Number : 3760003, Tel Litwinsky
- Italy (27):
  - Centro Sclerosi Multipla UO Neurologia Universitaria, Dipartimento di Neuroscienze, AOU S.Anna-Site Number : 3801025, Cona, Ferrara
  - Investigational Site Number : 3800008, Pozzilli, Isernia
  - Investigational Site Number : 3800016, Milan, Lombardy
  - Investigational Site Number : 3800032, Monza, Monza E Brianza
  - Investigational Site Number : 3800015, Rome, Roma
  - AOU S. Luigi Gonzaga-Site Number : 3801024, Orbassano, Torino
  - Investigational Site Number : 3801012, Catania
  - Investigational Site Number : 3800014, Chieti
  - Ospedale Valduce-Site Number : 3800033, Como
  - Investigational Site Number : 3801027, Cuneo
  - AOU CAREGGI-Site Number : 3800004, Florence
  - Policlinico "Riuniti" di Foggia-Site Number : 3800019, Foggia
  - Investigational Site Number : 3801011, Genova
  - Investigational Site Number : 3800002, Milan
  - A.O.U di Modena - Centro Sclerosi Multipla, Ospedale Civile di Baggiovara-Site Number : 3801028, Modena
  - A.O.U. Università degli studi della Campania Luigi Vanvitelli, II Clinica Neurologica-Site Number : 3801010, Napoli
  - AOU maggiore della carità di Novara-Site Number : 3801026, Novara
  - Investigational Site Number : 3801022, Palermo
  - Policlinico "P.Giaccone"U.O.C. di Neurologia - Centro Sclerosi Multipla-Site Number : 3800017, Palermo
  - Investigational Site Number : 3801029, Parma
  - Investigational Site Number : 3801005, Pavia
  - Investigational Site Number : 3801030, Ravenna
  - Investigational Site Number : 3800001, Roma
  - Investigational Site Number : 3801013, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Site Number : 3800021, Roma
  - Investigational Site Number : 3801031, Udine
  - Investigational Site Number : 3800020, Verona
- Japan (15):
  - Investigational Site Number : 3920002, Chiba, Chiba
  - Investigational Site Number : 3920013, Fukuoka, Fukuoka
  - Investigational Site Number : 3920003, Koriyama-shi, Fukushima
  - Investigational Site Number : 3920006, Asahikawa, Hokkaido
  - Investigational Site Number : 3920014, Asahikawa-shi, Hokkaido
  - Investigational Site Number : 3920017, Sapporo, Hokkaido
  - Investigational Site Number : 3920008, Morioka, Iwate
  - Investigational Site Number : 3920010, Sagamihara-shi, Kanagawa
  - Investigational Site Number : 3920001, Kyoto, Kyoto
  - Investigational Site Number : 3920015, Higashimatsuyama-shi, Saitama
  - Investigational Site Number : 3920016, Kodaira-shi, Tokyo
  - Investigational Site Number : 3920004, Meguro-ku, Tokyo
  - Investigational Site Number : 3920011, Ōta-ku, Tokyo
  - Investigational Site Number : 3920012, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920009, Tachikawa-shi, Tokyo
- Investigational Site Number : 4401001, Vilnius, Lithuania
- Investigational Site Number : 4581001, Kuala Lumpur, Malaysia
- Mexico (7):
  - Investigational Site Number : 4841007, Guadalajara, Jalisco
  - Investigational Site Number : 4841009, Delegacion Coyoacan, Mexico City
  - Investigational Site Number : 4840002, Monterrey, Nuevo León
  - Investigational Site Number : 4841005, Culiacán, Sinaloa
  - Investigational Site Number : 4840011, Yucatán, Yucatán
  - Investigational Site Number : 4841003, Tlalnepantla
  - Investigational Site Number : 4840001, Veracruz
- Poland (14):
  - Investigational Site Number : 6160002, Plewiska, Greater Poland Voivodeship
  - Investigational Site Number : 6160018, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6161005, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6161017, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6161008, Lodz, Lódzkie
  - Investigational Site Number : 6161016, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6161010, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160019, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6161011, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160004, Zabrze, Silesian Voivodeship
  - Investigational Site Number : 6160020, Żory, Silesian Voivodeship
  - Investigational Site Number : 6161014, Krakow
  - Investigational Site Number : 6160006, Rzeszów
  - Investigational Site Number : 6161015, Kielce, Świętokrzyskie Voivodeship
- Portugal (6):
  - Investigational Site Number : 6200001, Braga
  - Investigational Site Number : 6201005, Coimbra
  - Investigational Site Number : 6200009, Guimarães
  - Investigational Site Number : 6201011, Lisbon
  - Investigational Site Number : 6201012, Lisbon
  - Investigational Site Number : 6200002, Matosinhos Municipality
- San Juan MS Center- Site Number : 8401106, Guaynabo, Puerto Rico
- Romania (3):
  - Investigational Site Number : 6421004, Bucharest
  - Investigational Site Number : 6420002, Campulung Muscel
  - Investigational Site Number : 6421001, Constanța
- Investigational Site Number : 6820001, Riyadh, Saudi Arabia
- Investigational Site Number : 7021001, Singapore, Singapore
- Slovakia (4):
  - Investigational Site Number : 7031001, Bratislava
  - Investigational Site Number : 7030007, Martin
  - Investigational Site Number : 7030004, Nitra
  - Investigational Site Number : 7030003, Trnava
- South Africa (2):
  - Investigational Site Number : 7101002, Cape Town
  - Investigational Site Number : 7101001, Pretoria
- South Korea (7):
  - Investigational Site Number : 4100001, Goyang-si, Gyeonggi-do
  - Investigational Site Number : 4100007, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100008, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
- Spain (19):
  - Investigational Site Number : 7240007, Seville, Andalusia
  - Investigational Site Number : 7241016, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240010, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7241009, Barakaldo, Bizkaia
  - Investigational Site Number : 7241012, Donostia / San Sebastian, Gipuzkoa
  - Investigational Site Number : 7241024, Salt, Girona [Gerona]
  - Investigational Site Number : 7240013, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240001, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7241023, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7241022, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Córdoba
  - Investigational Site Number : 7240006, Madrid
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240005, Málaga
  - Investigational Site Number : 7240018, Murcia
  - Investigational Site Number : 7241008, Valencia
  - Investigational Site Number : 7240011, Valladolid
  - Investigational Site Number : 7241014, Vigo
- Investigational Site Number : 7561001, Bern, Switzerland
- Investigational Site Number : 1581001, Kaohsiung City, Taiwan
- Thailand (3):
  - Investigational Site Number : 7641002, Bangkok
  - Investigational Site Number : 7641001, Bangkok Noi
  - Investigational Site Number : 7641004, Khon Kaen
- Turkey (Türkiye) (19):
  - Investigational Site Number : 7921018, Ankara
  - Investigational Site Number : 7920011, Ankara
  - Investigational Site Number : 7921020, Bursa
  - Investigational Site Number : 7921013, Bursa
  - Investigational Site Number : 7921005, Eskişehir
  - Investigational Site Number : 7920012, Istanbul
  - Investigational Site Number : 7921016, Istanbul
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7921009, Istanbul
  - Investigational Site Number : 7920007, Istanbul
  - Investigational Site Number : 7921019, Izmir
  - Investigational Site Number : 7920008, Izmir
  - Investigational Site Number : 7921014, Kayseri
  - Investigational Site Number : 7920001, Kocaeli
  - Investigational Site Number : 7920015, Konya
  - Investigational Site Number : 7921006, Mersin
  - Investigational Site Number : 7921004, Samsun
  - Investigational Site Number : 7920017, Van
- Ukraine (9):
  - Investigational Site Number : 8040007, Chernivtsi
  - Investigational Site Number : 8040001, Chernivtsi
  - Investigational Site Number : 8040009, Ivano-Frankivsk
  - Investigational Site Number : 8041003, Ivano-Frankivsk
  - Investigational Site Number : 8041006, Kyiv
  - Investigational Site Number : 8040008, Lutsk
  - Investigational Site Number : 8040004, Lviv
  - Investigational Site Number : 8041002, Lviv
  - Investigational Site Number : 8041005, Vinnytsia
- United Kingdom (5):
  - Investigational Site Number : 8260001, Exeter, Devon
  - Investigational Site Number : 8261003, Canterbury, Kent
  - Investigational Site Number : 8260013, London, London, City of
  - Investigational Site Number : 8260010, Inverness
  - Investigational Site Number : 8261008, Salford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371
- See also: Multiple Sclerosis Website — https://www.sanofistudies.com/JQ2Z/
- See also: EFC17919 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25565&tenant=MT_SNY_9011